CLINICAL TRIAL: NCT06166810
Title: In Silico and in Vitro Targeting of Healthy Gut Bacteria With Fiber Degrading Metabolic Potential
Brief Title: Capture of Healthy Gut Bacteria Associated to High Fiber Diet
Acronym: iTARGET
Status: Recruiting | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-A01677-38
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-09

CONDITIONS: General Population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The role of the intestinal microbiota on health is now well recognised, and diet is one of the factors influencing the maintenance of a healthy intestinal microbiota. More specifically, the consumption of fruit, vegetables and cereals is associated with good health and, in particular, with an increase in the relative abundance of bacterial groups described as beneficial. To date, a large number of bacterial species in the intestinal microbiota have yet to be isolated and cultivated, which limits the characterisation of their potential health benefits. In order to isolate and cultivate these intestinal bacteria, it is particularly relevant to recruit individuals with a high-fibre diet.

DETAILED DESCRIPTION:
Since two decades, numerous studies have been performed to better understand the role of the gut microbiota in health and disease. An imbalance in the intestinal microbiota, known as dysbiosis, is frequently described as a cause of many chronic diseases and metabolic dysfunctions in humans. Among the factors that play an important role in maintaining this balance, diet plays a predominant role. More specifically, the consumption of fruit, vegetables and cereals is associated with good health and, in particular, with an increase in the relative abundance of bacterial groups described as beneficial. Modulating the intestinal microbiota via the or directly by providing these beneficial bacteria (next generation probiotics NGPs) is therefore a possible promising approach for the prevention and/or treatment of pathologies. To date, a large number of bacterial species in the intestinal microbiota have yet to be isolated and cultivated, which limits the characterization of their potential health benefits. Having strains that can be isolated and cultured is an essential step in phenotyping and characterization. In order to isolate and cultivate these intestinal bacteria, it is particularly important to recruit individuals with a high-fiber diet. In this context, a positive selection of donors, based on their dietary profiles highly enriched in fiber, is essential. In this study, the aim is to identify in silico unprecedented potentially new beneficial gut bacteria, and isolate, culture and characterize these bacterial species for their potential. This will be an innovative approach, using culturomics tools guided by metagenomics to isolate them. To do this, the fecal samples of 10 healthy volunteers will be collected with a regular and diversified intake of fruit, vegetables and cereals, which encourage the growth of beneficial micro-organisms and increase the richness of the intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects ;
* Age between 20 and 50 (limits included) ;
* BMI between 18.5 and 25 kg/m2 (excluding limits) ;
* Consumption of more than 5 portions of fruit and vegetables a day;
* Intake of at least 25g of dietary fibre per day;
* A varied diet with little processed food.

Exclusion Criteria:

* Antibiotics and/or transit modulators taken in the 3 months prior to sampling;
* Known pathologies;
* Current treatment;
* History of digestive surgery having an impact on the microbiota, deemed incompatible with the study (bariatric surgery);
* Consumption of food supplements based on protein preparations, probiotics or prebiotics;
* Smoking (even occasionally);
* Alcohol consumption > 2 glasses (i.e. 20 g) per day;
* Intense sporting activity;
* Pregnant or breast-feeding women;
* Persons under legal protection (curatorship, guardianship, etc.);
* Volunteers taking part in another intervention study;
* Persons refusing to be registered on the French Ministry of Health's Fichier National des Volontaires Sains (National Register of Healthy Volunteers);
* Subject not affiliated to the social security system;
* Subject in a period of exclusion from a previous study or having received a total amount of compensation exceeding 6000 euros over the 12 consecutive months prior to the start of the trial (after verification in the Fichier des Volontaires pour la Recherche Biomédicale).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: General population residing in Clermont-Ferrand (France)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Isolation and culture of one isolate from each target species | Up to 3 years
  Successful isolation and culture of at least one isolate from each target species previously identified through metagenomic data analyses.

SECONDARY OUTCOMES:
metagenomic profiles in relation to dietary profiles | Up to 3 years
  To obtain metagenomic profiles using shotgun sequencing of the gut microbiota (bacterial species), in relation to dietary profiles
growth capacity of the isolates | Up to 3 years
  To characterize the growth (growth monitoring by optical density) of the isolates of interest.
Functional potential of the isolates | up to 3 years.
  To characterize the genomic features of the isolates of interest (functional potential through genome annotation).
Phenotypic caracterization of the isolates | Up to 3 years
  To characterize phenotypically the isolates of interest by API gallery.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria MESLIER, PhD, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement; Claire CHERBUY, PhD, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- CRNH Auvergne, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No
No sharing planned

REFERENCES:
- [Derived] Caille A, Connan C, Lyon Belgy N, Borezee E, Cherbuy C, Meunier N, Meslier V. Positive nutritional selection of adults with healthy lifestyle and high daily fiber consumption for the isolation of beneficial intestinal bacteria: The iTARGET cohort study protocol. MethodsX. 2025 Mar 17;14:103268. doi: 10.1016/j.mex.2025.103268. eCollection 2025 Jun. PMID 40224142